CLINICAL TRIAL: NCT04150510
Title: Online Survey to Assess Smoking, Vaping, and Alcohol Consumption Behavior in the Population
Brief Title: Assessment of Smoking, Vaping, and Alcohol Consumption Behavior
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Professor; Director, Ingestive Behavior, Weight Management & Health Promotion Laboratory, Pennington Biomedical Research Center
Other Study IDs: 2019-052-PBRC
Record Dates: First submitted 2019-10-28; First posted 2019-11-04 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Survey; E-Cig Use; Smoking Behaviors; Alcohol Drinking; Vaping; Food Intake
MeSH Terms: conditions — Vaping; Smoking; Alcohol Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Online Survey: Individuals who are willing to participate in this online survey

SUMMARY:
To assess smoking, vaping, and alcohol consumption behaviors via online surveys in the population. Further, the objective is to administer additional surveys to assess which methods (e.g., pen-and-paper records, a smartphone app) for monitoring smoking, vaping, alcohol intake, and food intake are preferred by the study population.

DETAILED DESCRIPTION:
Many smokers believe that smoking helps them to control their weight, and concerns about weight gain can interfere with smoking cessation. In fact, nicotine has been shown to suppress appetite and increase resting metabolic rate, and smoking also serves as a behavioral alternative to eating or a distraction from hunger or food cravings. E-cigarettes are frequently marketed as the safer and healthier alternative to smoking, and some e-cigarettes are in fact actively advertised for weight management and/or suppression of food cravings, encouraging smokers to make the switch. In contrast, alcohol consumption has been shown to increase appetite and food intake and at the same time is associated with smoking and vaping.

Therefore, it is possible that participants who smoke or vape for weight control, particularly those who also regularly consume alcohol, would benefit from a lifestyle program that encompasses dietary counseling and exercise to prevent weight gain after smoking cessation. Additionally, methods to assess smoking, vaping, alcohol intake, and food intake (i.e., ingestive behaviors) historically relied on self-report, though the investigator's group has developed smartphone apps that allow people to capture images of their intake and/or self-report their intake in the app. App-based methods offer advantages, including the real-time transfer of data, and it is presumed that people will believe that apps are an easier and preferred method to capture ingestive behaviors, yet this assumption has not yet been thoroughly examined.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 85 years are eligible to complete the Demographics Questionnaire and the Food Intake Assessment Preference Questionnaire.
* Individuals in the same age range who regularly smoke cigarettes can complete the Smoking Questionnaire and the Smoking Assessment Preference Questionnaire, in addition to the Demographics Questionnaire and the Food Intake Assessment Preference Questionnaire
* Individuals in the same age range who regularly use e-cigarettes (vape) can complete the Vaping Questionnaire and the Vaping Assessment Preference Questionnaire, in addition to the Demographics Questionnaire and the Food Intake Assessment Preference Questionnaire
* Individuals in the same age range who regularly drink alcohol can complete the Alcohol Consumption Questionnaire and the Alcohol Consumption Assessment Preference Questionnaire, in addition to the Demographics Questionnaire and the Food Intake Assessment Preference Questionnaire

Individuals who engage in several of these behaviors can complete all questionnaires that apply.

Exclusion Criteria:

• Individuals who are unwilling to participate in this survey

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18 to 85 years who regularly engage in one or more of the following behaviors:
  * cigarette smoking
  * e-cigarette consumption (vaping)
  * alcohol consumption
Sampling Method: Non-Probability Sample
Enrollment: 3245 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Demographic data | Day of survey completion, up to 12 months
  age, sex, race/ethnicity, marital status, education, employment status, household income, zip code, height and weight, the prevalence of cardiovascular risk factors and cancer, and food security status
Smoking behavior | Day of survey completion, up to 12 months
  smoking status, history, frequency, amount, cues, motivation to quit, and potential factors affecting the decision to quit including the effect of smoking on food cravings
Vaping behavior | Day of survey completion, up to 12 months
  vaping status, history, frequency, amount, cues, motivation to quit and potential factors affecting the decision to quit including the effect of vaping on food cravings
Alcohol consumption | Day of survey completion, up to 12 months
  alcohol consumption status, history, frequency, amount, cues, motivation to quit/reduce consumption, and the effect of alcohol consumption on food cravings

SECONDARY OUTCOMES:
Smoking Assessment Preference | Day of survey completion, up to 12 months
  This questionnaire assesses the willingness to use different methods to monitor smoking behavior such as a pen-and-paper record or a smartphone app
Vaping Assessment Preference | Day of survey completion, up to 12 months
  This questionnaire assesses the willingness to use different methods to monitor vaping behavior such as a pen-and-paper record or diary, a 24-hour recall, or a smartphone app
Alcohol Consumption Assessment Preference | Day of survey completion, up to 12 months
  This questionnaire assesses the willingness to use different methods to monitor alcohol consumption such as a pen-and-paper record or diary, a 24-hour recall, or smartphone app-based methods (remote photography or in-app self-estimation of drink sizes)
Food Intake Assessment Preference Questionnaire | Day of survey completion, up to 12 months
  This questionnaire assesses the willingness to use different methods to monitor food intake such as a pen-and-paper record or diary, a 24-hour recall, or smartphone app-based methods (remote food photography or in-app self-estimation of portion sizes)

CONTACTS AND LOCATIONS:
Overall Officials: Corby K Martin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Access to individual de-identified data is possible via Pennington Biomedical Research Center's Data Sharing policy.